CLINICAL TRIAL: NCT04767620
Title: A Prospective, Open, Randomized, Controlled Phase Ⅱ Clinical Study of Ruxian Zengsheng No. 1 Decoction in Treating Liver-stagnation and Qi-stagnation Hyperplasia of Breast
Brief Title: Clinical Trial of Ruxian Zengsheng No. 1 Decoction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiuda Zhao (Other)
Responsible Party: Sponsor-Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Organization: Affiliated Hospital of Qinghai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHQU-2021002
Record Dates: First submitted 2021-02-09; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Mammary Gland Hyperplasia
Keywords: Mammary gland hyperplasia; Liver Qi stagnation

STUDY DESIGN:
Intervention Model Description: non
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study group took the No.1 Recipe for Rugden Zengsheng, and the control group took clinical observation and follow-up at the breast center. The study group and the control group were grouped randomly by envelope, and grouped according to 2:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study groups (Experimental): The study group was treated with Rugdenzengsheng No. 1 prescription for 2 courses.
  Interventions: Drug: Rugdenzengsheng No. 1 prescription
- control groups (No Intervention): The control group was treated with observational treatment and follow-up in outpatient clinic.

INTERVENTIONS:
Drug: Rugdenzengsheng No. 1 prescription — The study group was treated with the No. 1 Mammary Gland Growth Recipe orally, a total of 1 course of treatment, each course of 14 days, avoiding the menstrual period. The specific composition of Mammary Gland Hyperplasia No. 1 Recipe: Angelica 10g, Radix Paeoniae Alba 10g, Atractylodes Macrocephala 10g, Ginger 3g, Peppermint 6g, Vinegar Green Peel 6g, Lychee Seed 12g, Tangerine Seed 10g, Corydalis 10g, Fritillaria 6g, Trichosanthis 10g, Kombu 20g , Mustard seeds 10g, Moutan bark 6g, Poria 10g, North Bupleurum 6g. Method of administration: 14 doses in total, taken twice a day. The medicine is formulated in the herbal medicine room of the Affiliated Hospital of Qinghai University, with strict quality control.
  Other Names: non
  Arms: study groups

SUMMARY:
A prospective, open, randomized, controlled phase II clinical study is planned to clarify the efficacy and related adverse reactions of Mammary Glandular Hyperplasia No. 1 Decoction in the treatment of liver-qi stagnation type breast hyperplasia, relieve the pain of patients with breast hyperplasia, and improve the quality of life of patients.

DETAILED DESCRIPTION:
1. This study is a prospective, open, randomized, controlled Phase II clinical study. Strictly follow the design requirements of the clinical research, randomly enroll patients, control each link of the study with high quality, and obtain objective research results to improve the evidence-based medicine evidence of the breast hyperplasia treatment of liver-stagnation and qi stagnation type breast hyperplasia with Rugongshengsheng No.1 prescription;
2. Recruiting 137 patients with liver-stagnation and qi stagnation type breast hyperplasia through the Breast Center Clinic of the Affiliated Hospital of Qinghai University (see the inclusion criteria for details) (see the research plan for the specific calculation method), and randomly divided into 91 cases according to the 2:1 random number method Group, 46 cases of control group. The research group was treated with No.1 Rugdenzengsheng prescription for a total of 1 course of treatment, each course of 14 days, avoiding the menstrual period. The control group was given observation treatment and follow-up in outpatient clinic. All patients will be followed up by telephone or outpatient by a dedicated person, and the results of the follow-up will be recorded objectively;
3. Specific treatment plan: The study group was treated with Mammary gland Hyperplasia No. 1 orally, a total of 1 course of treatment, each course of 14 days, avoiding the menstrual period. The specific composition of Mammary Gland Hyperplasia No. 1 Recipe: Angelica 10g, Radix Paeoniae Alba 10g, Atractylodes Macrocephala 10g, Ginger 3g, Peppermint 6g, Vinegar Green Peel 6g, Lychee Seed 12g, Tangerine Seed 10g, Corydalis 10g, Fritillaria 6g, Trichosanthis 10g, Kombu 20g , Mustard seeds 10g, Moutan bark 6g, Poria 10g, Beibuihu 6g. Method of administration: 14 doses in total, taken twice a day. The medicine is formulated in the herbal medicine room of the Affiliated Hospital of Qinghai University, with strict quality control;
4. All patients will be followed up by telephone or on-site within one week after treatment. The evaluation criteria are detailed in the attached table. The curative effect evaluation standard of hyperplasia of mammary glands is mainly through the scoring method. The analgesic curative effect standard (NRS score on the most painful day): clinical recovery: the pain disappears completely; marked effect: the pain is significantly reduced, only occasional pain or only slight tenderness; effective : Pain is reduced or tenderness is reduced; Ineffective: Pain remains unchanged or worsened. In addition, collect clinical pathological data of patients, such as age, gender, reproductive history, menstrual history, family history, breastfeeding history, etc.;
5. Secondary efficacy indicators: safety evaluation, safety endpoints include the incidence of adverse events and adverse reactions, liver function, renal function and urine routine laboratory examinations before and after treatment;
6. Apply for ethical review by the ethics committee of the Affiliated Hospital of Qinghai University, and conduct research in strict accordance with the ethical requirements of the ethics committee of the Affiliated Hospital of Qinghai University.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women over 18 years of age;
2. Patients who meet the diagnostic criteria for breast color Doppler ultrasound diagnosis of breast hyperplasia and the course of disease exceeds 3 months;
3. Meet the syndrome differentiation criteria for liver-stagnation and qi stagnation (main symptoms are ① breast distension Pain and pain; ② breast pain and/or lumps are related to menstruation and mood changes; ③ irritability and irritability; ④ flank fullness. Secondary symptoms: ① the lumps are single, soft and tender; ② Young women; ③Irregular menstruation or dysmenorrhea; ④Pale red tongue, thin white or thin yellow coating, stringy pulse. With 3 main symptoms or 2 main symptoms + 2 secondary symptoms);
4. breast color ultrasound, breast molybdenum Target, or breast MRI showed BI-RADS 2-3;
5. NRS (0-10 pain rating) score ≥ 4 points on the most painful day before treatment, according to the score, the pain is divided into mild 3 points, moderate Grade 4-6 points, severe 7-10 points;
6. Voluntarily participate in the clinical study and sign the informed consent form after the informed consent (patients voluntarily accept the study and sign the informed consent).

Exclusion Criteria:

1. Patients with other breast diseases or other causes of breast pain (such as mastitis, breast cancer, etc.);
2. Patients with severe cardiovascular and cerebrovascular diseases, liver, kidney, malignant tumors, blood system diseases, and Patients with mental illness;
3. Patients who have been confirmed to have dysfunctional uterine bleeding, amenorrhea, polycystic ovary syndrome, menopausal syndrome and hyperprolactinemia before treatment, still need to regulate hormone levels for treatment;
4. Patients diagnosed with hypercortisolism before treatment still need bromocriptine treatment;
5. Menstrual period is more than 7 days, menopause and severe irregular menstrual cycle;
6. ALT, AST, ALP, TBIL , GGT is higher than the upper limit of normal; or abnormal blood, urine, electrocardiogram and other examination items;
7. pregnant or breastfeeding women, or patients with pregnancy plans in the next six months;
8. 1 before treatment Use Chinese or Western medicine to treat breast hyperplasia (including painkillers, topical drugs, acupuncture, etc.) within the month and during the treatment period, and use hormonal drugs (except for long-term use), and oral contraceptives within six months;
9. People who are known to be allergic to the ingredients of the test drug prescription;
10. Past alcohol or drug abuse history;
11. Patients who participated in other clinical studies within 3 months before enrollment;
12. According to the judgment of the researchers, there are other diseases Or circumstances will reduce the possibility of enrollment or complicate enrollment. For example, frequent changes in the work environment may cause loss to follow-up, and patients with mental and behavioral disorders, or the inability to sign informed consent.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult healthy women over 18
Enrollment: 137 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Relief Rate of Mammary Gland Pain | 12 weeks
  To clarify the effectiveness of Rugshengsheng No.1 Recipe in the Affiliated Hospital of Qinghai University in reducing the pain of patients with liver-stagnation and qi stagnation type breast hyperplasia, as well as related adverse side effects, and provide reliable clinical evidence for further clinical promotion

SECONDARY OUTCOMES:
Relief time of breast pain | 12 weeks
  Related Adverse Reactions of Rugongshengsheng No.1 Prescription
Related adverse reactions | 12 weeks
  Statistic about the related adverse reactions of patients after taking the No.1 Recipe for Mammary Gland Growth, the degree and severity of the adverse reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Qinghai, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: No